CLINICAL TRIAL: NCT03227939
Title: Effect of Laparoscopic Sleeve Gastrectomy (LSG) Plus Uvulopalatopharyngoplasty and Adenoidectomy/Tonsillectomy on Severe Obstructive Sleep Apnea & Hyponea Syndromes in Moderate-to-severe Obese Patients: an Open-label Randomized Controlled Clinical Trial
Brief Title: Effects of Combined Surgery on Obstructive Sleep Apnea in Obese Patients: an Open-label Randomized Controlled Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bing Wang (Other)
Responsible Party: Sponsor-Investigator, Bing Wang, Professor of Surgery, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Organization: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JYLJ013
Record Dates: First submitted 2017-07-20; First posted 2017-07-24 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: To Compare the Difference of AHI Variation Between LSG and Combined Surgery
MeSH Terms: interventions — Adenoidectomy; Tonsillectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined Surgery Group (Experimental): LSG + UPPP＆Adenoidectomy/Tonsillectomy
  Interventions: Procedure: Laparoscopic sleeve gastrectomy（LSG）; Procedure: Uvulopalatopharyngoplasty(UPPP) and Adenoidectomy/Tonsillectomy
- LSG Group (Active Comparator): LSG only
  Interventions: Procedure: Laparoscopic sleeve gastrectomy（LSG）

INTERVENTIONS:
Procedure: Laparoscopic sleeve gastrectomy（LSG） — LSG：All these operations were performed by the same surgeon team. Dissect the greater omentum alongside the greater gastric curvature, make sure that the greater gastric curvature and fundus of stomach were completely made free from pancreas and spleen.Fully Exposed left and right diaphragm angle and taking care not to injure the esophagus. Resection was started 2 to 4 cm from pylorus and alongside a 40Fr tube up to the esophagogastric junction and created a 60 to 80ml gastric lumen, removed the fundus of stomach thoroughly and take care of the esophagus and preventriculus. Repaired the hiatal hernia if it was exsit.
Procedure: Uvulopalatopharyngoplasty(UPPP) and Adenoidectomy/Tonsillectomy — UPPP：PPP is typically administered to patients with obstructive sleep apnea in isolation. It is administered as a stand-alone procedure in the hope that the tissue which obstructs the patient's airway is localized in the back of the throat. The rationale is that, by removing the tissue, the patient's airway will be wider and breathing will become easier.
  Arms: Combined Surgery Group

SUMMARY:
This research is created for compare the difference of AHI variation between LSG and combined surgery on obstructive sleep apnea in obese patients , evaluate the risk of combined surgery and explore the correlative factor of the curative effect.

DETAILED DESCRIPTION:
Obesity is one of the new health challenges in China and all over the world，Morbidly obesity (MO) is an important risk factor for metabolic diseases and obstructive sleep apnea(OSA), which can be effectively and lastingly reduced by bariatric surgery.

OSA is the most common type of sleep apnea and is caused by complete or partial obstructions of the upper airway. It is characterized by repetitive episodes of shallow or paused breathing during sleep, and is a potentially fatal disease. OSA has complex pathogenesis and numerous pathogeny, while morbidly obesity is one of the important risk factors of OSA. Previous research has shown that the incidence of OSA will rise by 1.14 % while body mass index(BMI) rise by 1%.Therefor, loseing weight is highly recommend for morbidly obese patients with OSA in clinical guideline for OSA both in USA and China, and bariatric surgery is effective for morbidly obese patients with OSA. Most yellow race morbidly obesity patients have abdominal obesity which is different from the white race，while Abdominal obesity is associated with greater incidence and more severely of OSA. There are maybe twenty million patients with OSA and 80% of them haven't been diagnosed.

At present,. Laparoscopic sleeve gastrectomy(LSG) and laparoscopic Roux-en-Y gastric bypass(LRYGB) are two of the main bariatric surgical procedures performed in China. They can performed as one stage each or multiple sessions(LSG-LRYGB) which is depend on the severity of obesity and its complications.

UPPP was first performed in 1981 by doctor Fujita and modified these years, it has been a standardized treatment for OSA. The effective rate of UPPP is less than 65% and is associated with the BMI and age of patients , younger and lower BMI means better effect. Consideration of the discontented outcome in obese patients, Simple UPPP is not recommended for OSA patients with morbidly obesity in clinical guidelines for OSA.

Although simple LSG has a sure prostecdtive efficacy for both OSA and morbidly obesity, patients still need CPAP during several months after surgery. So we chosed patients who conformed the surgical indications of both morbidly obesity and OSA，and performed an combined surgery (LSG+UPPP+adenoidectomy/tonsillectomy). We found that combined surgery has a better short-term efficacy than simple LSG, so the randomized clinical trial(RCT) was designed to explore the efficacy of combined surgery in the treatment of severe OSA in moderate-to-severe obese patients.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese Han population aged 16 to 65 years
2. BMI more than 32.5Kg/㎡ with AHI more than ≥30/hour
3. First diagnosed with PSG without any corresponding treatment;
4. Adenoid tonsil hypertrophy (Friedman stage II-III).

Exclusion Criteria:

1. Drug abuse, alcohol addiction and mental diseases
2. Dysgnosia
3. Over-high expectation
4. Risk-averse patient;
5. Poor tolerance to surgery
6. Patient suffering from gastroesophageal reflux and hiatal hernia
7. Central or mixed sleep apnea diagnosed by PSG
8. PO2<60mmHg when the patient is awake
9. Suffering from maligent tumor, neural system injury and respiratory insufficiency
10. Hypothyroidism
11. Other special issue decided by specialist.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-07-25 (Estimated); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
The mean change in Apnoea-Hypopnoea Index (AHI) | At the 6 month after surgery
  The mean change in AHI

SECONDARY OUTCOMES:
Time to response | during 6 months after surgery
  AHI reduse to 50% of the base line
Other PSG measures: average and lowest blood oxygen saturation at night | At the 6 month after surgery
  in psg report
Weight, BMI | At the 6 month after surgery
neck,chest,waist hip and biceps circumference | At the 6 month after surgery
Epworth Sleepiness Scale (ESS) scores | At the 6 month after surgery
Changes in the CT scan of upper airway and head radiography | At the 6 month after surgery

IPD SHARING:
Plan to Share IPD: Undecided